CLINICAL TRIAL: NCT02110849
Title: Longitudinal Study for the Evaluation of Safety and Efficacy Parameters in Prostate Cancer Patients Treated at IU Health Proton Therapy Center (IUHPTC)
Brief Title: Prostate Cancer Parameters for Patients Receiving Proton Treatment
Status: Withdrawn | Type: Observational
Why Stopped: Closure of IU Health Proton Facility
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: IUHPTC-03; IRB #1206008885 (Other: Indiana University)
Record Dates: First submitted 2014-04-03; First posted 2014-04-10 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: Prostate; Proton Therapy; Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Protons

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prostate Cancer Patients: Prostate cancer patients who received proton radiation therapy
  Interventions: Radiation: Proton

INTERVENTIONS:
Radiation: Proton — Proton Therapy for Prostate Cancer

SUMMARY:
To prospectively collect data from patients treated with proton therapy for prostate cancer using the IUHPTC technique for the evaluation of toxicity and efficacy of this treatment technique.

DETAILED DESCRIPTION:
The major purpose of this study is to analyze side effects experienced and self-reported by prostate cancer patients undergoing proton radiation therapy at IUHPTC. With the information collected, the investigators will establish pre-existing conditions before proton treatment and measure side effects after treatments that are not related to the pre-existing conditions. Also, to compare long-term side effects for patients who are treated with hormone suppression therapy along with their proton therapy to those patients who do not get treated with hormone suppression therapy. This information will help doctors better understand the side effects experienced and may help provide valuable information for future patients making decisions regarding their treatment options.

Finally, to develop a database of information regarding the treatment and outcomes for patients with prostate cancer in order to improve care of patients with this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed adenocarcinoma of the prostate and are scheduled to receive proton radiation treatment at IUHPTC.
* Subjects with any stage or grade of tumor will be allowed including proton salvage therapy in the context of a rising PSA after surgery and a negative metastatic work-up.
* Prior use of Lupron therapy or a similar agent is allowed. Use of Lupron or similar agent must be for ≤ 6 months prior to enrollment.
* Use of Casodex and agents in the same drug class is allowed. Age is ≥ 18 years at the time of consent.
* The ability to understand and willingness to sign an informed consent and authorization for the release of health information.

Exclusion Criteria:

-Evidence of distant metastases at the time of enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients who are receiving proton radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
To prospectively collect a composite of toxicity events on patients who treated with proton therapy for prostate cancer using the IUHPTC technique for the evaluation of toxicity and efficacy of this treatment technique. | 12 months
  A collection of toxicity events of proton therapy, evaluate the long-term side effects of hormone suppression vs. non-hormone suppression and documents the clinical benefits this therapy in regards to urinary, sexual and gastrointestinal issues.
  To do this the investigators will use the following standard of care data collection forms that include; the International Index of Erectile Function (Attachment 1), the American Urological Association Symptom Index (Attachment 2) and the Radiation Therapy Initial Nursing Assessment (Attachment 3), The prostate preexisting conditions review (attachment 4) and the prostate side effects review (attachment 5). Other clinical data such us demographics, vitals, previous treatments, PSA(prostate specific antigen/Hormone results, follow up data, as described in the protocol schedule of events, will be collected as per routine standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Buchsbaum, MD, Principal Investigator — Indiana University Proton Therapy Center
Locations (1):
- Iu Health Proton Therapy Center, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No data collected